CLINICAL TRIAL: NCT03248037
Title: Randomized, Double-masked, Placebo-controlled Evaluation of Netarsudil for Prevention of Corticosteroid-induced Intraocular Pressure Elevation
Brief Title: Trial of Netarsudil for Prevention of Corticosteroid-induced Intraocular Pressure Elevation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cornea Research Foundation of America (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2017-003
Record Dates: First submitted 2017-08-09; First posted 2017-08-14 (Actual); Results first posted 2021-02-12 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-01

CONDITIONS: Fuchs' Endothelial Dystrophy; Bullous Keratopathy
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy | interventions — netarsudil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Netarsudil (Experimental): Netarsudil ophthalmic solution 0.02%, dosed topically once a day for 9 months
  Interventions: Drug: Netarsudil
- Placebo (Placebo Comparator): Placebo eye drop, dosed topically once a day for 9 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Netarsudil — netarsudil opthalmic solution 0.02%
  Arms: Netarsudil
Drug: Placebo — Placebo eye drops
  Arms: Placebo

SUMMARY:
Cornea transplant recipients who are using topical corticosteroids long-term to prevent transplant rejection will be randomized to use netarsudil or placebo.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age; male or female patient undergoing Descemet membrane endothelial keratoplasty; patient is able and willing to administer eye drops; patient is able to comprehend and has signed the Informed Consent form; patient is likely to complete the nine-month course of the study.

Exclusion Criteria:

* A patient exhibiting pre-operative intraocular inflammation; a patient with a known sensitivity to any of the ingredients in the study medications; a patient who has a condition (i.e., UNCONTROLLED systemic disease) or is in a situation which in the investigator's opinion may put the patient at significant risk, may confound the study results, or may interfere significantly with the patient's participation in the study; a patient with abnormal eyelid function; a patient that is exhibiting active corneal ulceration, keratitis, or conjunctivitis, or who has a history of herpetic keratitis; a patient who has been diagnosed with uncontrolled glaucoma, prior aqueous shunt or trabeculectomy, or with preoperative intraocular pressure > 22 mm Hg in the potential study eye; presence of any ocular disease that would interfere with the evaluation of the study treatment (however, patients with a history of cystoid macular edema, age-related macular degeneration, corneal neovascularization, and other non-interfering comorbidities may be enrolled); a patient with a history of non-compliance with using prescribed medication; a patient who is concurrently involved in or participated in another randomized clinical trial within 30 days prior to enrollment in this study; patients who are pregnant or planning to become pregnant within the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2019-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis W Price, Jr, MD, Principal Investigator — Price Vision Group
Locations (1):
- Price Vision Group, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fini ME, Schwartz SG, Gao X, Jeong S, Patel N, Itakura T, Price MO, Price FW Jr, Varma R, Stamer WD. Steroid-induced ocular hypertension/glaucoma: Focus on pharmacogenomics and implications for precision medicine. Prog Retin Eye Res. 2017 Jan;56:58-83. doi: 10.1016/j.preteyeres.2016.09.003. Epub 2016 Sep 22. PMID 27666015
- [Background] Vajaranant TS, Price MO, Price FW, Gao W, Wilensky JT, Edward DP. Visual acuity and intraocular pressure after Descemet's stripping endothelial keratoplasty in eyes with and without preexisting glaucoma. Ophthalmology. 2009 Sep;116(9):1644-50. doi: 10.1016/j.ophtha.2009.05.034. Epub 2009 Jul 29. PMID 19643499
- [Derived] Price MO, Feng MT, Price FW Jr. Randomized, Double-Masked Trial of Netarsudil 0.02% Ophthalmic Solution for Prevention of Corticosteroid-Induced Ocular Hypertension. Am J Ophthalmol. 2021 Feb;222:382-387. doi: 10.1016/j.ajo.2020.09.050. Epub 2020 Oct 10. PMID 33045216

RESULTS

PARTICIPANT FLOW:
Recruitment Details: As specified in the protocol, a total of 120 unique participants were enrolled in the study; 71 enrolled both eyes in the study and the fellow eyes were automatically assigned to opposite treatment arms, so 71 subjects participated in both treatment arms.
Units Other Than Participants: eyes
Period: Overall Study
Arm/Group | Netarsudil | Placebo
Started | 95; 95 eyes (Fellow eyes could be enrolled and were automatically assigned to the opposite treatment arm.) | 96; 96 eyes (Fellow eyes could be enrolled and were automatically assigned to the opposite treatment arm.)
Completed | 74; 74 eyes | 87; 87 eyes
Not Completed | 21; 21 eyes | 9; 9 eyes
Not completed — Withdrawal by Subject | 6 | 9
Not completed — Adverse Event | 15 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Netarsudil | Placebo | Total
Number analyzed (Participants) | 95 | 96 | 191
Age, Continuous [Median (Full Range); unit: years] | 68 [40 to 88] | 67 [40 to 90] | 67 [40 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 61 | 115
  Male | 41 | 35 | 76
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 95 | 96 | 191

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure
Description: Intraocular pressure measurement exceeding 24 mm Hg or more than 10 mm Hg greater than the pre-randomization reading.
Time Frame: from date of randomization until the date of first documented intraocular pressure elevation exceeding defined threshold up to 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Netarsudil | Placebo
Number analyzed (Participants) | 95 | 96
Participants | 11 | 18

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Netarsudil | Placebo
All-Cause Mortality (participants affected / at risk) | 0/95 | 0/96
Serious Adverse Events (participants affected / at risk) | 0/95 | 0/96
Other Adverse Events (participants affected / at risk) | 31/95 | 18/96
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Netarsudil (N=95) | Placebo (N=96)
Air re-injection (Eye disorders) | 20 (20) | 18 (18) — Air was re-injected into the eye to promote endothelial keratoplasty attachment
Ocular irritation considered related to study drug use (Eye disorders) | 22 (22) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-23): https://cdn.clinicaltrials.gov/large-docs/37/NCT03248037/Prot_SAP_000.pdf